CLINICAL TRIAL: NCT04359212
Title: Increased Risk of Venous Thromboembolism and Higher Hypercoagulable State in Patients Recovered in Intensive Care Unit and in Medical Ward for Coronavirus Disease 2019 (COVID-19)
Brief Title: Increased Risk of VTE and Higher Hypercoagulability in Patients Recovered in ICU and in Medical Ward for COVID-19
Acronym: VTE-COVID
Status: Completed | Type: Observational
Sponsor: Quovadis Associazione (Other)
Collaborators: Azienda Ospedaliera di Padova (Other)
Responsible Party: Sponsor
Other Study IDs: VTE-COVID
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-04

CONDITIONS: COVID-19 Disease; Thromboembolism, Venous
Keywords: COVID-19 pandemic; Thromboembolism, Venous; Deep Venous Thrombosis; Pulmonary Thrombosis
MeSH Terms: conditions — Venous Thromboembolism; COVID-19; Venous Thrombosis | interventions — Heparin, Low-Molecular-Weight; Fondaparinux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical: subject with a confirmed infection for COVID-19 and needing admission to a medical division for a non-severe clinical disease
  Interventions: Drug: thromboprophylaxis with low-molecular-weight heparin or fondaparinux
- Intensive: subject with a confirmed infection for COVID-19 and needing admission to an Intensive Cure Unit for a severe to critical disease
  Interventions: Drug: thromboprophylaxis with low-molecular-weight heparin or fondaparinux

INTERVENTIONS:
Drug: thromboprophylaxis with low-molecular-weight heparin or fondaparinux — thromboprophylaxis with low-molecular-weight heparin or fondaparinux
  Other Names: thromboprophylaxis

SUMMARY:
The aim of this study is to verify if patients admitted to hospital in a medical division and in the intensive care unit for a COVID-19 infection are at higher risk of developing a VTE complication and if they actually present an increased hypercoagulable state.

DETAILED DESCRIPTION:
Between December 2019 and January 2020, a new type of coronavirus, named as "coronavirus disease 2019 - COVID-19" by the World Health Organization, has widely spread throughout the world, becoming a global health threat. The new COVID-19 is similar to other two types of coronavirus that in the past two decades have emerged as cause of severe human disease: Severe Acute Respiratory Syndrome CoV (SARS-CoV) and Middle East Respiratory Syndrome CoV (MERS-CoV). Severe respiratory disease or respiratory failure are the principal symptoms of critical patients, needing a management in ICU with mechanical ventilation.18 Data coming from laboratory results show a leucopenia mainly represented by a lymphopenia, that is a cardinal feature of COVID-19. Moreover, the concentration of several serum pro-thrombotic cytokines, such as interleukins (mainly IL-6, increased in 52% of patients), TNF-α, D-Dimer are reported to be significantly higher in COVID-19 patients, and significantly higher in ICU-patients than in non-ICU patients, suggesting an increased hypercoagulable state that, joined to the other main risk factors (immobilization, ICU admission, mechanical ventilation, infective disease), place these patients to a potential greater risk of developing VTE complications.

ELIGIBILITY:
Inclusion Criteria:

* aged >= 18 years
* needing admission to a medical hospital division or to an ICU
* with a confirmed infection for COVID-19

Exclusion Criteria:

* aged < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients aged > 18 years with a confirmed infection for COVID-19 and needing admission to a medical division for a non-severe clinical disease (Group 1) or to the ICU for a severe to critical disease (Group 2) will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
the cumulative proportion of any distal or proximal deep venous thrombosis or of symptomatic pulmonary embolism | 28 days
  the cumulative proportion of any distal or proximal deep venous thrombosis or of symptomatic pulmonary embolism

SECONDARY OUTCOMES:
the cumulative proportion of any distal or proximal deep venous thrombosis or of symptomatic pulmonary embolism plus the asymptomatic incidentally detected pulmonary embolism | 28 days
  the cumulative proportion of any distal or proximal deep venous thrombosis or of symptomatic pulmonary embolism plus the asymptomatic incidentally detected pulmonary embolism

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Simioni, MD, Principal Investigator — Department of Medicine, University of Padua (I)
Locations (1):
- Giuseppe Camporese, Padua, Italy

REFERENCES:
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Flumignan RL, Tinoco JDS, Pascoal PI, Areias LL, Cossi MS, Fernandes MI, Costa IK, Souza L, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Prophylactic anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD013739. doi: 10.1002/14651858.CD013739. PMID 33502773